CLINICAL TRIAL: NCT06578910
Title: Retrospective, Non-interventional Clinical Investigation of the Safety and Performance of 640AD Monofocal Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Medicontur Medical Engineering Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: M_640AD_HU_2204
Record Dates: First submitted 2024-06-10; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Cataract; Pseudophakia
Keywords: Intraocular lens; Ametropia - correction; Presbyopia- correction
MeSH Terms: conditions — Cataract; Pseudophakia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 640AD: 80 patients (105 eyes) implanted with 640AD IOL monocularly or binocularly
  Interventions: Diagnostic Test: Standard of care; Other: Patient satisfaction questionnare

INTERVENTIONS:
Diagnostic Test: Standard of care — 12 months after the IOL implantation: measurement of intraocular pressure, slitlamp and fundus examination, visual acuity, manifest refraction.
Other: Patient satisfaction questionnare — VFQ- 25 (Visual Function Questionnare) to be completed during 12 month visit.

SUMMARY:
Medicontur hydrophilic posterior chamber monofocal intraocular lens (IOL) is indicated to improve vision at far distance in adults with cataract and/or ametropia (hyperopia, myopia), secondarily to removal of the crystalline lens.

The intraocular lens is intended to be surgically implanted into the eye with the purpose of restoring optical function in the aphakic eye to provide an optical system with high predictability of the precalculated dioptric power.

The study will be performed partially as a retrospective study with patients enrolled who had been implanted with 640AD IOLs mono- or binocularly between December 2021 - December 2022.

Data from five visits will be collected:

* Baseline preoperative (maximum 30 days prior to surgery)- retrospective
* IOL implantation Day 0 - retrospective
* Postoperative visit at Day 1 (+/- 0 days) - retrospective
* Postoperative visit at 1 month (+/- 2 weeks) - retrospective
* Postoperative visit at 12 months (+/- 3 months) - consent and prospective visit

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females above 18 years of age;
* Pseudophakic patients implanted with 640AD monofocal IOLs (implanted between December 2021 - December 2022);
* Diagnosis of cataract and/or ametropia (hyperopia, myopia);
* Subject who has signed an informed consent form.
* Patients who have participated in all visits that are subject to retrospective data collection.

Exclusion Criteria:

* Patients who are not targeted to emmetropia ( outside -0,5 and 0,5 D)
* Patients with the following condition(s) at the time of the baseline visit:

  * Corneal astigmatism > 1.5 D
  * Uncontrolled diabetic retinopathy
  * Iris neovascularization
  * Congenital eye abnormality
  * Uncontrolled glaucoma
  * Pseudoexfoliation syndrome
  * Amblyopia
  * Uveitis
  * AMD (advanced AMD)
  * Retinal detachment
  * Prior ocular surgery in personal medical history
  * Previous laser treatment
  * Corneal diseases
  * Severe retinal diseases (dystrophy, degeneration)
  * High myopia
  * Inadequate visualization of the fundus on preoperative examination
  * Patients deemed by the clinical investigator because of any systemic disease
  * Pregnancy
  * Eye trauma in medical history
  * Current use of systemic steroids or topical ocular medication
* Patients with any eye condition that could affect vision in the opinion of the investigator at the time of the 12-month follow-up: (corneal ectasia, retinal diseases, glaucoma, uveitis, dry eye or amblyopia, etc.)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults (18 years old and older) with cataract and/or ametropia (hyperopia, myopia), who have undergone monocular or binocular implantation with the 640AD IOL model.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Monocular corrected distance visual acuity (CDVA) | 12 months postoperatively
  To compare monocular corrected distance visual acuity (CDVA) between 12 months postoperative and preoperative results.

SECONDARY OUTCOMES:
Monocular uncorrected distance visual acuity (UDVA) | 12 months postoperatively
  To compare monocular uncorrected distance visual acuity (UDVA) at 12 months postoperative and preoperative status.
UDVA and CDVA | 12 months postoperatively
  To compare percentage of eyes that achieve monocular UDVA and monocular CDVA within logMAR 0.0 or 0.3 at 12 months postoperative and preoperative status.
Manifest residual refraction | 12 months postoperatively
  To compare residual SPH at 12 months postoperative and preoperative status. (Residual CYL and axis are not applicable, as it is a monofocal IOL, that does not correct astigmatism)
Patient satisfaction | 12 months postoperatively
  Visual Function Questionnaire 25 (National Eye Institute) is used to evaluate overall satisfaction, subjective perception of colour perception and scotopic vision at 12 months postoperatively. The results are evaluated according to the official evaluation guide.

OTHER OUTCOMES:
Safety outcome - Intraoperative complications | Day1 postoperatively
  Intraoperative complications of cataract surgery
  * Posterior capsular or zonular rupture
  * Vitreous loss/anterior vitrectomy or aspiration
  * Iris/ciliary body injury
  * Loss of nuclear material into vitreous
  * Suprachoroidal haemorrhage
  * Retrobulbar haemorrhage
Safety outcome - Postoperative complications | Month1 postoperatively
  Postoperative complications of cataract surgery
  * Cystoid macular oedema
  * Iris abnormalities
  * Corneal oedema
  * Wound leak or rupture
  * IOL dislocation, removal, or exchange
  * Inflammation (Endophthalmitis, anterior chamber cells, anterior chamber flare, hypopyon)
  * Retinal tear, break, or detachment
  * Persistent iritis
  * Elevated intraocular pressure
  * Pupillary block
  * Cornea status
Safety outcome - Complications of IOL implantation | Month12 postoperatively
  Complications of IOL implantation
  * Posterior capsular opacification (PCO)
  * Opacification, IOL discoloration

CONTACTS AND LOCATIONS:
Locations (1):
- SZTE ÁOK Szent-Györgyi Albert Klinikai Központ Szemészeti Klinika, Szeged, Hungary